CLINICAL TRIAL: NCT00973167
Title: The Efficacy of Low-magnitude, High-frequency Vibration Treatment on Reducing Fracture Risks and Fracture Incidences in the Community Elderly - a Prospective Randomized Trial
Brief Title: Low-magnitude High-frequency Vibration Study on Fracture Rate in Community Elderly
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kwok-Sui Leung, Chair Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 469508
Record Dates: First submitted 2009-08-05; First posted 2009-09-09 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Fractures
Keywords: Fracture rate; Fracture risks
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Remains sedentary with normal lifestyle
- Treatment (Experimental): Receive LMHFV treatment for 18 months.
  Interventions: Device: Low-magnitude high-frequency vibration treatment

INTERVENTIONS:
Device: Low-magnitude high-frequency vibration treatment — Stand on a vibration platform at 35Hz, 0.3g, 20mins/day and 5 days/week
  Arms: Treatment

SUMMARY:
Fragility fracture is common due to global aging problem, incurring huge healthcare expenditure. The occurrence of fragility fracture is usually caused by a fall incidence of an elderly with low bone quality and poor balancing ability. Therefore, any approach to improve or retard both sarcopenia and osteoporosis will be helpful to prevent osteoporotic fracture incidence. With the intensive research on low magnitude high frequency vibration (LMHFV), many scientific evidences support the application of this biophysical modality on elderly to maintain or improve the musculoskeletal tissues in elderly.

Many previous studies showed the osteogenic properties of vibration treatment and its positive effects on muscular performance and blood circulation. The investigators' previous reports also indicated that LMHFV could enhance the bone quality in spine and tibia in elderly after one-year intervention, as well as the balancing ability with high compliance. In animal studies, the application of LMHFV on fracture healing also demonstrated the significant acceleration of healing by inducing callus formation and maturation, from which upregulation of collagen I, II and BMP-2 gene expression was detected at molecular level. To date, the long-term efficacy of LMHFV on reducing fracture risks and fracture rate is, however, not available, which needs a systematic large-scale study to answer this important research question.

Therefore, the hypothesis of this study is that LMHFV can maintain or enhance the performance of various tissues of the musculoskeletal system in community elderly, thus reducing the fracture risks and fracture rate. A large-scale prospective randomized clinical trial will be conducted in multiple communities to investigate the long-term effect of LMHFV on fracture rate and reduction of fracture risks in community elderly, in which multi-factorial effects, in terms of muscle and bone, on musculoskeletal system will also be evaluated. A total of 704 elderly from 28 community centres will be recruited within 1.5-year time for a 18-month LMHFV treatment, who will be assessed on the fracture risks at fixed time points while their fracture rates on the third year of this study will be regarded as primary outcome for analysis. The findings of this study will provide very useful scientific data to support the application of LMHFV for elderly. The ultimate goal is to reduce the fracture rate and the quality of life of community-living elderly.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or above
* independent in accessing the centres

Exclusion Criteria:

* having habitual exercise or participate in supervised exercise
* having drug treatment that affects normal metabolism of musculoskeletal system
* having hypo- or hyperparathyroidism, renal, liver or other chronic diseases
* having low-energy fracture history
* previous or current smokers or drinkers

Ages: 65 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 704 (Actual)
Dates: Start 2009-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Fracture rate | up to 18 months

SECONDARY OUTCOMES:
Balancing ability | up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Kwok-Sui Leung, MD, Principal Investigator — Department of Orthopaedics & Traumatology, The Chinese University of Hong Kong
Locations (1):
- Department of Orthopaedics & Traumatology, The Chinese University of Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Leung KS, Li CY, Tse YK, Choy TK, Leung PC, Hung VW, Chan SY, Leung AH, Cheung WH. Effects of 18-month low-magnitude high-frequency vibration on fall rate and fracture risks in 710 community elderly--a cluster-randomized controlled trial. Osteoporos Int. 2014 Jun;25(6):1785-95. doi: 10.1007/s00198-014-2693-6. Epub 2014 Mar 28. PMID 24676848